CLINICAL TRIAL: NCT01614665
Title: A Phase II, Parallel Group, Randomized, Multicentre, Open Label Study to Compare the Pharmacokinetics of Tacrolimus in De Novo Pediatric Allograft Recipients Treated With an Advagraf® or Prograf® Based Immunosuppressive Regimen, Including a Long-Term Follow-Up
Brief Title: A Study to Compare How the Body Absorbs and Processes Two Different Formulations of the Anti-rejection Medication Tacrolimus (Advagraf® or Prograf®) in Children Receiving an Organ Transplant, and How Safe and Effective They Are Over a Longer Period of Time
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PMR-EC-1207; 2011-000078-80 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplantation; Kidney Transplantation; Liver Transplantation
Keywords: Transplant; Prograf; Heart; Advagraf; Tacrolimus; Immunosuppression; Kidney; Liver; Pharmacokinetic; Pediatric
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): Participants receive tacrolimus twice daily starting from day 1 for 4 weeks for in Part A, and continue to receive tacrolimus twice daily up to end of Part B and C of the study.
  Interventions: Drug: Tacrolimus
- Tacrolimus Prolonged Release (Experimental): Participants receive tacrolimus prolonged release once daily starting from day 1 for 4 weeks for in Part A, and continue to receive tacrolimus prolonged release once daily up to end of Part B and of the study.
  Interventions: Drug: Tacrolimus prolonged release

INTERVENTIONS:
Drug: Tacrolimus — Participants receive an initial total daily dose of tacrolimus depending on the type of organ transplant (heart = 0.075 mg/kg; liver/kidney = 0.3 mg/kg), to be given orally (or via nasogastric tube for liver transplant recipients) in 2 doses in the morning and the evening. The first dose is administered in the morning within days of skin closure (heart = 4 days; liver = 2 days; kidney = within 24 hours following reperfusion). Subsequent tacrolimus doses are taken orally twice a day in the morning and evening and are adjusted on the basis of clinical evidence of efficacy, occurrence of adverse events and observing the recommended whole blood trough level ranges (day 1 through 21 = 10 to 20 ng/mL; day 22 through 365 = 5 to 15 ng/mL).
  Other Names: Prograf; FK506
  Arms: Tacrolimus
Drug: Tacrolimus prolonged release — Participants receive an initial total daily dose of tacrolimus prolonged release depending on the type of organ transplant (heart = 0.075 mg/kg; liver/kidney = 0.3 mg/kg), to be given orally (or via nasogastric tube for liver transplant recipients) in 1 dose. The first dose is administered in the morning within days of skin closure (heart = 4 days; liver = 2 days; kidney = within 24 hours following reperfusion). Subsequent tacrolimus prolonged release doses are taken orally once a day in the morning and are adjusted on the basis of clinical evidence of efficacy, occurrence of adverse events and observing the recommended whole blood trough level ranges (day 1 through 21 = 10 to 20 ng/mL; day 22 through 365 = 5 to 15 ng/mL).
  Other Names: Prograf XL; Graceptor; FK506 (MR4); Advagraf; Astagraf XL
  Arms: Tacrolimus Prolonged Release

SUMMARY:
The purpose of this study is to compare how the body absorbs and processes two different formulations of the anti-rejection medication tacrolimus (Advagraf® or Prograf®) in children receiving an organ transplant, and how safe and effective they are over a longer period of time.

This study is for children less than 16 years old. No minimum age has been set, however, to be included in this study participants must able to swallow the medication capsules intact.

DETAILED DESCRIPTION:
Participants undergoing primary heart, kidney or liver transplantation and meeting the Inclusion Criteria and complying with the Exclusion Criteria prior to initiation of tacrolimus therapy will be enrolled.

Participants will be randomized to treatment with either Advagraf® or Prograf®. The randomization will be on a 1:1 basis stratified by organ and centre.

The study is divided in to two parts:

Part A: The initial pharmacokinetic part of the study.

Part B: A long term follow-up of one year. The main objective of Part A of the study is to collect PK data following administration of Advagraf® and Prograf® in de novo pediatric allograft recipients. Part B allows comparison of the safety and efficacy profiles of Advagraf® vs. Prograf® for longer term (52 weeks) post allograft transplantation.

Part C: Continuation of long-term follow-up (from Day 365 onwards). Participants who have completed Part B and to whom continued treatment with Advagraf® is not currently available, will be offered participation in a continuation of long-term follow-up Part C. Part C will continue until Advagraf® becomes available to these participants or these participants' discontinuation, whichever is the earliest.

This applies to participants in the following countries: Czech Republic, Italy, UK and Poland only.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged <16 years of age, undergoing primary liver, kidney or heart allograft transplantation
* The subject must be able to swallow intact Prograf® or Advagraf® capsules
* Subjects, treated since transplantation with Basiliximab or ATG/ Mycophenolate Mofetil (MMF)/steroids, whose gastric motility has resumed and whose renal function is adequate on Day 1 (Heart only)

Exclusion Criteria:

* Subject is receiving a multi-organ transplant or has previously received an organ transplant (including re-transplantation)
* Subject with pulmonary vascular resistance ≥4 Wood units despite medication
* Subject with significant renal impairment, defined as having serum creatinine ≥230 μmol/l (≥2.6 mg/dl) pre-transplantation. (Not applicable for renal transplanted subjects)
* Subject with significant liver disease, defined as having continuously elevated SGPT/ALT and/or SGOT/AST and/or total bilirubin levels of ≥3 times the upper value of the normal range of the investigational site during the past 28 days. (Not applicable for liver transplanted subjects)
* Subject with malignancies or a history of malignancy within the last 5 years, with the exception of those with basalioma or squamous cell carcinoma of the skin that has been treated successfully. (Not applicable for transplanted subjects with a primary organ diagnosis of cancer)
* Subject requiring systemic immunosuppressive medication for any other indication than transplantation

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2012-04-03 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve from Time 0 to Time 24 Hours (AUC0-24h) for Tacrolimus (Part A) | Days 1, 7 and 28 at predose, 1, 2, 4, 6, 12, 13, 14, 16, 18 and 24 hours postdose
Number of Participants with Adverse Events (Part A + B) | From first dose of study drug up to 7 days after last dose of study drug in Part B (up to 53 weeks)
  Safety is assessed by adverse events (AEs), which includes abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induces clinical signs or symptoms, needs active intervention, interruption or discontinuation of study medication or is clinically significant. A serious AE (SAE) is an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, is life-threatening, requires or prolongs hospitalization or is considered medically important.
Number of Participants with Adverse Events (Part C) | Up to 9 years
  Safety is assessed by adverse events (AEs), which includes abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induces clinical signs or symptoms, needs active intervention, interruption or discontinuation of study medication or is clinically significant. A serious AE (SAE) is an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, is life-threatening, requires or prolongs hospitalization or is considered medically important.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of Tacrolimus (Part A) | Days 1, 7 and 28 at predose, 1, 2, 4, 6, 12, 13, 14, 16, 18 and 24 hours postdose
Time to Attain Maximum Concentration (tmax) of Tacrolimus (Part A) | Days 1, 7 and 28 at predose, 1, 2, 4, 6, 12, 13, 14, 16, 18 and 24 hours postdose
Trough Concentration (C12) for Tacrolimus (Part A) | Days 1, 7 and 28, 12 hours after dosing
Trough Concentration (C24) for Tacrolimus (Part A) | Days 1, 7 and 28, 24 hours after dosing
Correlation between AUC24 & C24 (Part A) | Days 1, 7 and 28 at predose, 1, 2, 4, 6, 12, 13, 14, 16, 18 and 24 hours postdose
Number of Participants with Acute Rejections (Part A + B) | Up to Week 52
  Rejection episodes/acute rejections are indicated by clinical and/or laboratory signs, and are classified according to their rejection specific treatment: •Spontaneously Resolving Acute Rejection: not treated with new or increased corticosteroid medication, antibodies or any other medication and resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Sensitive Acute Rejection: treated with new or increased corticosteroid medication only and which has resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Resistant Acute Rejection: did not resolve following treatment with corticosteroids; - Resolved with further treatment: any acute rejection with an end date AND a treatment other than corticosteroid used; - Unresolved with further treatment: any acute rejection with no end date AND a treatment other than corticosteroid used; - Unresolved with no further treatment: any acute rejection with no end date AND ONLY corticosteroid treatment was used.
Number of Participants with Biopsy-proven Acute Rejection Episodes (BPARs) (Part A + B) | Up to Week 52
  BPAR episodes are defined as acute rejection episodes confirmed by biopsy, and are classified according to their rejection specific treatment: •Spontaneously Resolving Acute Rejection: not treated with new or increased corticosteroid medication, antibodies or any other medication and resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Sensitive Acute Rejection: treated with new or increased corticosteroid medication only and which has resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Resistant Acute Rejection: did not resolve following treatment with corticosteroids; - Resolved with further treatment: any acute rejection with an end date AND a treatment other than corticosteroid used; - Unresolved with further treatment: any acute rejection with no end date AND a treatment other than corticosteroid used; - Unresolved with no further treatment: any acute rejection with no end date AND ONLY corticosteroid treatment used.
Severity of Biopsy Proven Acute Rejection Episodes (Part A + B) | Up to Week 52
  The severity of BPARs is categorized with specific criteria by organ: For kidney transplant participants, according to Banff '97 Diagnostic categories for renal allograft biopsies - Banff '07 update (C4d deposition, Acute antibody-mediated rejection I, II, and III, Acute T cell mediated rejection IA, IB, IIA, IIB and III); for liver transplant participants, according to 1997 Banff Schema for Grading of Liver Allograft Rejection - Rejection Activity Index (mild, moderate, severe or indeterminate/borderline); for heart, according to Standardized Nomenclature of the International Society of Heart and Lung Transplantation - Standardised Cardiac Biopsy Grading: Acute Cellular Rejection 2004 (mild, moderate, severe).
Patient Survival (Part A + B) | Up to Week 52
  Patient survival is defined as the time from first dose of study drug to the date of death from any cause.
Graft Survival (Part A + B) | Up to Week 52
  Graft survival is defined as the time from the first dose of study drug to graft loss. Graft loss is defined as retransplantation, nephrectomy (in case of kidney transplantation), death or dialysis (in case of kidney transplantation) ongoing at end of study or at discontinuation, unless superseded by follow-up information.
Efficacy Failure (Part A + B) | Up to Week 52
  Efficacy failure is defined as the composite of the following: death, graft loss, BPAR and unknown outcome. A participant is considered to have an unknown outcome if he/she does not have the event of interest (death, graft loss, BPAR) or does not have a study assessment prior to day 335.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe Ltd.
Locations (10):
- Site CZ61, Prague, Czechia
- France (2):
  - Site FR33, Bron
  - Site FR32, Paris
- Site IT52, Rome, Italy
- Site PL71, Warsaw, Poland
- United Kingdom (5):
  - Site GB43, Birmingham
  - Site GB46, Liverpool
  - Site GB44, London
  - Site GB45, London
  - Site GB42, Manchester

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/PMR-EC-1207/
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14383&tenant=MT_AST_9011